CLINICAL TRIAL: NCT00562432
Title: A Randomized Study to Demonstrate the Safety and Feasibility of Plexisyl-AF Administered to the Epicardial Fat Pads in Patients Undergoing Open-chest Coronary Artery Bypass Grafting (CABG)
Brief Title: A Randomized Study to Demonstrate the Safety and Feasibility of Plexisyl-AF in Patients Undergoing Coronary Artery Bypass Grafting (CABG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LoneStar Heart, Inc. (Industry)
Responsible Party: Andy Hinson, VP Clinical & Regulatory Affairs, LoneStar Heart, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYM-07-001; EudraCT Number 2007-006728-37
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2008-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; CABG; ganglionated plexi
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plexisyl-AF (Experimental): Plexisyl-AF implants
  Interventions: Device: Plexisyl-AF
- No Treatment (Sham Comparator): Surgery without experimental treatment
  Interventions: Device: Plexisyl-AF; Other: No Treatment

INTERVENTIONS:
Device: Plexisyl-AF — Plexisyl-AF implants
  Other Names: Standard surgery without device
Other: No Treatment — CABG without the experimental treatment
  Other Names: surgery without device
  Arms: No Treatment

SUMMARY:
The primary goal of this study is to assess the safety of Plexisyl-AF administered by direct application to the cardiac fat pads in patients undergoing coronary artery bypass grafting. Secondary goals of the study are to assess the potential response of Plexisyl-AF to reduce the occurrence of postoperative atrial fibrillation and assess the performance of the electrostimulator device to confirm the location of the epicardial fat pads (nerves). The occurrence of postoperative atrial fibrillation will be monitored by continuous cardiac monitoring.

DETAILED DESCRIPTION:
The purpose of this study is to investigate a non-surgical and non-destructive approach to providing a temporary, protective parasympathectomy as a means to reducing postoperative atrial fibrillation following cardiac surgery. Applications of Plexisyl-AF will be placed in the cardiac fat pads as a means for creating a "non-destructive" cardiac denervation.

This is a randomized assessment to demonstrate the safety of Plexisyl-AF in patients undergoing open heart surgery. Eligible patients will be those submitted to undergo open-chest CABG. Patients will receive Plexisyl-AF, administered via direct application to the SA nodal and AV nodal epicardial fat pads during the surgical procedure.

Patients will be monitored for the occurrence of atrial fibrillation via the use of continuous cardiac monitoring for a period of 120 hours following surgery. Patients will return the clinic for brief follow-up, including electrocardiographic recordings, 10 days, 30 days and 90 days after the date of surgery.

ELIGIBILITY:
Inclusion Criteria

1. The patients must be able and willing to give written informed consent.
2. The patients will be adult (age ≥ 18 years and </= 70 years) males or females who are scheduled to undergo on-pump open-chest coronary artery bypass grafting surgery of two (2) or more arteries.
3. The patients should be effectively treated prior to enrollment with an appropriate medical regimen (such as aspirin, ß-blockers, nitrates, and ACE inhibitors). Changes to medications after enrollment should be avoided.
4. If female, the patients must be (a) post-menopausal, (b) surgically sterile or (c) using adequate birth control and have a negative pregnancy test within 7 days prior to administration of device.

Exclusion Criteria

1. Emergent open heart surgery.
2. Patients scheduled to undergo mitral valve surgery, aortic, pulmonic or tricuspid valve replacements, and replacement or reconstruction of the aorta.
3. Patients who have undergone a previous open chest CABG procedure.
4. Previous history of atrial fibrillation or flutter.
5. Patient with clinical hypothyroidism or hyperthyroidism.
6. Prophylactic medication for the prevention of atrial fibrillation or current use of an antiarrhythmic medication. Patients who have been receiving beta-blockers and calcium channel blockers before screening may continue taking the medication.
7. First-degree or higher degrees of atrioventricular (AV) block (PR interval >210 msec)
8. An ejection fraction of less than 30%.
9. Clinically active congestive heart failure.
10. Serum creatinine > 2.0 mg/dL or currently receiving dialysis.
11. Clinically significant liver enzyme abnormalities (i.e., AST or ALT more than two times the upper limit of normal and/or bilirubin more than 50% above the upper limit of normal).
12. The patients will not be receiving concurrently an investigational product in another clinical trial or have received an investigational product in another clinical trial in the 30 days prior to enrollment.
13. Any other condition that, in the opinion of the clinical investigator, might compromise any aspect of the trial.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Plexisyl-AF administered by direct injection to the epicardial fat pads, evaluated through analysis of freedom from adverse experiences, clinical laboratory tests, electrocardiogram and physical examinations. | 90 days

SECONDARY OUTCOMES:
freedom from atrial fibrillation | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bauernschmitt, MD, Principal Investigator — Munich Heart Center
Locations (3):
- Germany (3):
  - Heart Center Dresden, Dresden
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, Munich